CLINICAL TRIAL: NCT02436915
Title: The Effects of Noninvasive Brain Stimulation on Physical and Mental Functioning in Older Adults
Acronym: BrainSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); The Falk Medical Research Trust, Bank of America, N.A. Trustee (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-002
Record Dates: First submitted 2015-04-10; First posted 2015-05-07 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2018-01

CONDITIONS: Aging
Keywords: Slow gait; Executive function; Transcranial direct current stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real tDCS (Experimental): The "real tDCS" intervention will consist of 10 daily 20-minute sessions of transcranial direct current stimulation (tDCS) targeting left prefrontal cortex at a target current intensity of 1.5 mA.
  Interventions: Other: Real tDCS
- Sham tDCS (Sham Comparator): The "sham tDCS" intervention will consist of 10 daily 20-minute sessions of transcranial direct current stimulation with same montage as the "real tDCS", except current will only be applied for the first 60 seconds of each session.
  Interventions: Other: Sham tDCS

INTERVENTIONS:
Other: Real tDCS — Transcranial direct current stimulation (tDCS) enables noninvasive, selective and sustained modulation of cortical activation. tDCS works by sending low-level currents between two or more scalp electrodes, which alters brain polarity and thus, perfusion and cortical excitability.
  Arms: Real tDCS
Other: Sham tDCS — For sham tDCS, current will only be applied for the first 60 seconds of each 20 minute session. This is a reliable sham control as sensations arising from tDCS diminish considerably after the first minute of stimulation.
  Arms: Sham tDCS

SUMMARY:
The objective of this study is to determine whether augmentation of prefrontal brain excitability using noninvasive transcranial direct current stimulation (tDCS) lessens the severity of the symptom triad associated with cerebral microvascular disease (CMD); that is, slow gait, cognitive dysfunction and depressive symptoms. Investigators will complete this objective by conducting a pilot, double-blinded randomized controlled trial of a 10-day intervention of real versus sham tDCS in 40 subjects.

DETAILED DESCRIPTION:
Biological aging, especially when coupled with cardiovascular risk factors, leads to chronic endothelial dysfunction within cerebral micro-vessels that impairs the brain's ability to meet the metabolic demands placed upon it by everyday life. This chronic mismatch between blood supply and metabolic demand often leads to cerebral microvascular disease (CMD), or the accumulation of ischemic damage within a network of frontal and subcortical regions. CMD is recognized as white matter hyperintensities on MRI scans and manifests clinically as mobility impairment, executive dysfunction and depressed affect. As 11-17% of elderly individuals present with this constellation of symptoms, and each of these symptoms is independently linked to increased morbidity and mortality, CMD is a critical yet understudied healthcare issue with rapidly-growing personal and economic costs.

There is currently no cure for CMD and trials aimed at pharmacological improvement of nonselective systemic vasodilation report no therapeutic value (Sorrond & Lipsitz, 2011). Our team, however, has demonstrated that the severity of clinical symptoms suffered by those with CMD is critically dependent upon the brain's remaining capacity to activate the appropriate cortical networks when metabolic demand is increased by the performance of various cognitive-motor tasks (Purkayastha et al., 2014; Sorond et al., 2010; Sorond et al., 2011). Therefore, investigators predict that improvement in the capacity to activate the appropriate cortical networks in response to increased metabolic demand would ameliorate the symptoms and improve the quality of life of patients with CMD.

Transcranial direct current stimulation (tDCS) enables noninvasive, selective and sustained modulation of cortical activation. tDCS works by sending low-level currents between two or more scalp electrodes, which alters brain polarity and thus, perfusion and cortical excitability. One 20-minute session of tDCS targeting the left prefrontal cortex acutely increases cortical activation during both cognitive and motor task performance in healthy adults. Investigators have demonstrated that this same stimulation improves mobility and cognitive performance in community-dwelling older adults. Moreover, repeated tDCS sessions over a one month period reduce symptoms of depression and may improve executive function in healthy individuals. This preliminary evidence suggests that tDCS may be an effective intervention for CMD; however, the impact of tDCS on this disease has not been investigated.

The study investigators ultimately aim to investigate the therapeutic efficacy of tDCS in patients with CMD by conducting a double-blind, proof-of-principle, sham-controlled trail along with extensive functional and neurophysiological assessments. In order to finalize the design and plan the implementation of this definitive trial, investigators currently aim to:

1. Conduct a pilot study to establish the feasibility of deployment of tDCS in large populations of individuals with CMD, and to obtain preliminary evidence for a causal effect of the intervention on mobility, executive function and depressive symptoms in this population.
2. Within the pilot study, investigate the effects of the tDCS intervention on cortical activation in response to cognitive-motor tasks.

This study will provide first-of-its-kind, proof-of-principle evidence on whether tDCS provides meaningful symptomatic relief to patients with CMD. Moreover, it will inform a more definitive, larger-scale randomized controlled trial (RCT) by providing information on recruitment and retention, compliance, estimates of effect size, and the neurophysiological underpinnings of expected functional improvements. If successful, knowledge gained is also expected to spur the investigation of tDCS as treatment for many other diseases-from dementia to diabetes-that negatively impact the brain's capacity to activate appropriate cortical networks.

ELIGIBILITY:
Inclusion Criteria:

* Slow gait, defined by an over-ground preferred walking speed of less than or equal to 1.0 m/s.
* Executive dysfunction, defined by a Trail Making Test B z-score of greater than one standard deviation below age- and gender-based norms.

Exclusion Criteria:

* Non-ambulatory
* Clinical history or brain imaging evidence of a previous stroke
* Parkinson's Disease
* Normal pressure hydrocephalus
* Other neurodegenerative condition
* Severe depression
* Lower-extremity arthritis or pain causing slow gait
* Inability or unwillingness to understand or participate in the study protocol
* Contraindications to MRI or tDCS, including (but not limited to) personal or family history of epilepsy, use of neuro-active drugs, claustrophobia or risk of metal objects in the body.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hebrew Rehabilitation Center, Roslindale, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Real tDCS: The "real tDCS" intervention will consist of 10 daily 20-minute sessions of transcranial direct current stimulation (tDCS) at a target current intensity of 1.5 mA.
  Real tDCS: Transcranial direct current stimulation (tDCS) enables noninvasive, selective and sustained modulation of cortical activation. tDCS works by sending low-level currents between two or more scalp electrodes, which alters brain polarity and thus, perfusion and cortical excitability.
- Sham tDCS: The "sham tDCS" intervention will consist of 10 daily 20-minute sessions of transcranial direct current stimulation, except current will only be applied for the first 60 seconds of each session.
  Sham tDCS: For sham tDCS, current will only be applied for the first 60 seconds of each 20 minute session. This is a reliable sham control as sensations arising from tDCS diminish considerably after the first minute of stimulation.
Period: Overall Study
Arm/Group | Real tDCS | Sham tDCS
Started | 9 | 10
Completed | 9 | 9
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real tDCS | Sham tDCS | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.10 (10.36) | 78.12 (10.79) | 80.46 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.17 (4.44) | 31.46 (5.75) | 30.38 (5.15)
Gait Speed [Mean (Standard Deviation); unit: m/s] | 0.73 (0.17) | 0.73 (0.14) | 0.73 (0.15)
Difference between the time to complete Trail Make Test Section B section and Section A [Mean (Standard Deviation); unit: seconds] | 148.62 (81.64) | 143.57 (71.96) | 145.94 (74.24)
Geriatric Depression Scale Score [Mean (Standard Deviation); unit: units on a scale] — Geriatric Depression Scale Score ranges from 0 to 15. greater score means greater depression. The score greater than 5 is considered as depression.
  units on a scale | 3.00 (3.02) | 4.00 (2.55) | 3.06 (2.21)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Post Intervention on Mobility
Description: Mobility and turning will be assessed by the timed up-and-go test (TUG) (Podsiadlo & Richardson, 1991). The participant will be seated in an armed chair. On the word "go," the subject will stand up using the arm rests if needed, walk (with assistive device if needed) around a cone placed three meters in front of the chair, return and sit down as quickly as possible. Time to complete the TUG test will be used as the outcome measure.
Time Frame: baseline, immediately after intervention and 2 weeks post intervention
Population: 19 participants were enrolled in the study and completed baseline assessments. One participant withdrew from the follow-up session due to illness deemed unrelated to participation. 18 participants completed all the study sessions.
Measure: Mean (Standard Deviation); unit: percent change of TUG time
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
percent change of TUG time
  Percent Change (Baseline to Immediate Follow Up) | -3.0 (17.1) | 10.4 (37.2)
  Percent Change (Baseline to 2-Week Follow up) | -6.1 (17.6) | 3.4 (24.1)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Equivalence — We hypothesized that the real tDCS would improve the performance of TUG (i.e., greater percent decrease of time to complete TUG from baseline to follow ups) as compared to the sham tDCS; p = 0.24, ANOVA

2. Primary Outcome: Percent Change From Baseline to Post Intervention on Global Cognition Impairment
Description: The Montreal Cognitive Assessment (MoCA) score is used as the outcome measure of Global Cognition Impairment. MoCA score ranges from 0 to 30. Lower MoCA score represents poorer cognitive function (i.e., more severe Global Cognition Impairment).
Time Frame: Baseline, immediately after intervention and 2 weeks post intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
percent change
  Percent Change (Baseline to Immediate Follow Up) | 7.9 (16.9) | 0.1 (8.2)
  Percent Change (Baseline to 2-Week Follow up) | 12.6 (14.5) | -0.4 (7.8)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Equivalence — We hypothesized that the real tDCS would improve the MoCA score (i.e., greater percent increase decrease of MoCA score from baseline to follow ups) as compared to the sham tDCS; p = 0.03, ANOVA

3. Primary Outcome: Percent Change From Baseline to Post Intervention on Dual Task Cost to Walking Speed in 24-meter Walking Test
Description: Six 24-meter walking trials at a preferred speed are completed and each three of them are in normal or dual task condition. The GaitRite pressure mat (Havertown, PA) will be used to record bilateral foot placements and measure the walking speed. Dual task cost to walking speed is defined as the percent change of walking speed from normal walking to dual task walking. The outcome was calculated by averaging the dual task costs of the six trials.
Time Frame: baseline, immediately after intervention and 2 weeks post intervention
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
percent change
  Percent Change (Baseline to Immediate Follow Up) | 14.9 (17.3) | 3.9 (14.5)
  Percent Change (Baseline to 2-Week Follow up) | 6.1 (8.4) | 3.9 (14.5)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Equivalence — We hypothesized that the real tDCS would improve the dual task performance of walking (i.e., greater percent decrease of dual task cost to walking speed from baseline to follow ups) as compared to the sham tDCS; p = 0.37, ANOVA

4. Primary Outcome: Percent Change From Baseline to Post Intervention on Dual Task Cost to Standing Postural Sway Speed
Description: Postural sway speed - assessed by measuring standing postural sway (ie., center-of pressure fluctuations) during six, 30-second trials of standing with eyes open (single task) or performing a cognitive task (dual task standing) on a stationary force platform (Kistler, Amherst, NY). Dual task cost is defined as the percent change of sway speed from single task standing to dual task standing. The outcome was obtained by averaging the dual task costs of the six trials.
Time Frame: baseline, immediately after intervention and 2 weeks post intervention
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
percentage change
  Percent Change (Baseline to Immediate Follow Up) | -23.1 (24.5) | 16.5 (27.5)
  Percent Change (Baseline to 2-Week Follow up) | -11.5 (20.2) | 15.3 (30.6)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Equivalence — We hypothesized that the real tDCS would improve the performance of dual task standing (i.e., greater percent decrease of dual task cost to standing sway speed from baseline to follow ups) as compared to the sham tDCS; p = 0.004, ANOVA

5. Secondary Outcome: Percent Change From Baseline to Post Intervention on Geriatric Depression Scale (GDS) Score
Description: GDS total Score. The GDS total score ranges from 0 to 15. Higher GDS score represents more severe depression.
Time Frame: baseline, immediately after intervention and 2 weeks post intervention
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
percent change
  Percent Change (Baseline to Immediate Follow Up) | 10.5 (54.4) | -12.9 (72.6)
  Percent Change (Baseline to 2-Week Follow up) | 27.3 (92.5) | -2.4 (76.2)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Equivalence — We hypothesized that the real tDCS would reduce the depression (i.e., greater percent decrease of GDS score from baseline to follow ups) as compared to the sham tDCS; p = 0.37, ANOVA

6. Secondary Outcome: Percent Change From Baseline to Post Intervention on Trial Making Test (TMT)
Description: Time to complete Trail Making Test part B minus time to complete TMT part A. Slower time to complete TMT-B as compared to TMT-A represents poorer executive function.
Time Frame: baseline, immediately after intervention and 2 weeks post intervention
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
percent change
  Percent Change (Baseline to Immediate Follow Up) | -65.8 (25.2) | -17.1 (49.5)
  Percent Change (Baseline to 2-Week Follow up) | -38.1 (34.8) | -17.2 (58.9)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Equivalence — We hypothesized that the real tDCS would improve the performance of TMT (i.e., greater percent decrease of time to complete TMT from baseline to follow ups) as compared to the sham tDCS; p = 0.54, ANOVA

7. Secondary Outcome: Percent Change From Baseline to Post Intervention on Dual-task Cost to Standing Sway Area
Description: Postural sway speed - assessed by measuring standing postural sway (ie., center-of pressure fluctuations) during six, 30-second trials of standing with eyes open (single task) or performing a cognitive task (dual task standing) on a stationary force platform (Kistler, Amherst, NY). Dual task cost is defined as the percent change of sway area from single task standing to dual task standing. The outcome was calculated by averaging the dual task costs of the six trials.
Time Frame: baseline, immediately after intervention and 2 weeks post intervention
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
percentage change
  Percent Change (Baseline to Immediate Follow Up) | -32.9 (43.6) | 51.1 (54.2)
  Percent Change (Baseline to 2-Week Follow up) | -34.4 (24.3) | 211.8 (153.2)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Equivalence — We hypothesized that the real tDCS would improve the performance of dual task standing (i.e., greater percent decrease of dual task cost to standing postural sway area from baseline to follow ups) as compared to the sham tDCS; p = 0.0007, ANOVA

8. Secondary Outcome: Percent Change From Baseline to Post Intervention on Dual Task Cost to Stride Time in 24-meter Walking Test
Description: Six 24-meter walking trials at a preferred speed are completed and each three of them are in normal or dual task condition. The GaitRite pressure mat (Havertown, PA) will be used to record bilateral foot placements and measure the walking speed. Dual task cost to stride time is defined as the percent change of stride time from normal walking to dual task walking.The outcome was calculated by averaging the dual task costs of the six trials.
Time Frame: baseline, immediately after intervention and 2 weeks post intervention
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
percent change
  Percent Change (Baseline to Immediate Follow Up) | -25.7 (38.4) | 83.8 (175.5)
  Percent Change (Baseline to 2-Week Follow up) | -16.3 (37.1) | 57.0 (136.9)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Equivalence — We hypothesized that the real tDCS would improve the performance of walking (i.e., greater percent decrease of dual task cost to stride time from baseline to follow ups) as compared to the sham tDCS; p = 0.04, ANOVA

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Real tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 1/8 | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real tDCS (N=8) | Sham tDCS (N=9)
Injurious Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — No hospitalization required, unrelated to study intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No